CLINICAL TRIAL: NCT04495582
Title: Observational Study of Long-term Safety and Efficacy of Subjects Who Participated in CS10BR05 Inj. Phase 1 Study
Brief Title: Long-term Follow-up of Phase 1 Clinical Trial of CS10BR05(CS10BR05-MSA101)
Status: Completed | Type: Observational
Sponsor: Corestemchemon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS10BR05-MSA101-E
Record Dates: First submitted 2020-07-21; First posted 2020-08-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Multiple System Atrophy
Keywords: Mesenchymal stem cell; Cell therapy; Multiple system atrophy; Neuroprotection; CS10BR05; Long-term Safety Study
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Interventional Study group: Subjects participating in this observational study originally participated in CS10BR05 Inj. phase 1 study.

SUMMARY:
The study purpose is conducting follow-up surveillance for the incidence of adverse events and efficacy of subjects participated in phase 1 trial to evaluate the safety and tolerability of autologous bone marrow-derived mesenchymal stem cells (CS10BR05) in subjects with Multiple System Atrophy until 60 months from administering investigational product (IP).

DETAILED DESCRIPTION:
Multiple system atrophy is a neurodegenerative disease of the central nervous system which is accompanied by signs of autonomic imbalance (orthostatic hypotension, urinary problems and erectile dysfunction), Parkinson's symptoms (movement decreases and limb tremors) and cerebellar ataxia symptoms (grogginess and incorrect pronunciation). It shows signs similar to Parkinson's disease, however, it doesn't show improvement of symptoms by dopaminergic drugs and occurs at any age.

The purpose is conducting follow-up surveillance for the incidence of adverse events and efficacy of subjects participated in phase 1 trial to evaluate the safety and tolerability of autologous bone marrow-derived mesenchymal stem cells (CS10BR05) in subjects with Multiple System Atrophy until 60 months from administering investigational product (IP).

Because it is the following observational study for subjects participated in phase 1 trial, there is no additional administration of the investigational product in the study.

If the subjects who participated in phase 1 trial voluntarily consent in writing to take part in this observational study, the subjects visit the institution according to the protocol that designed the follow-up visits every 3 months (Visit 1, Visit 2) until 6 months from administration of investigational product and since then 6 months later (Visit 3), every 12 months (Visit 4~7) to observe the incidence of adverse events and efficacy.

As a result of evaluating severity of AE divided into subjective, objective in accordance with the CTCAE (Version 4.0) standards.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the phase 1 clinical trial(Protocol No.: CS10BR05- MSA101) at 3 months after administering investigational product
* Subjects who give a written, signed and dated informed consent spontaneously

Exclusion Criteria:

* Subjects who decided as inappropriate cases to participate in the observational study by investigator

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The subjects who participated in the phase 1 clinical trial(NCT03265444, Protocol No.: CS10BR05-MSA101) will be enrolled in this study, so the number of enrolled subjects will depend on the number of actual enrolled subjects for the phase 1 clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Safety assessment(evaluation) | 5 years
  1. Adverse events(AE): After the completion of the CS10BR05-MSA101 phase 1 trial, new adverse events, including tumor are assessed and detailed information is collected at each visit. Whole body PET test is performed for tumor observation at visit 7.
  2. Laboratory test: The following laboratory tests are performed at each visit.
     * Hematology test: WBC, RBC, Hemoglobin, Hematocrit, Platelets count, WBC Diffcount
     * Chemistry test: Na, K, Ca, Cl, BUN, Creatinine, Uric acid, Total bilirubin, Albumin, Total protein, Creatine Kinase, Cystatin-C, ALT, AST, r-GT, ALP, LDH, Glucose, Total cholesterol, Triglyceride
     * Urine test: Protein, Glucose, Urobilinogen, WBC, RBC
  3. Measuring vital signs (blood pressure in mmHg, heart rate in bpm, body temperature in Celsius) is performed at each visit.
  4. Physical examination is performed at each visit. If clinically significant abnormal findings are recorded in the CRF and collected as AEs.
Efficacy assessment(evaluation) | 5 years
  The following tests are conducted at each visit to exploratively evaluate the efficacy. Evaluate the change of score of each tools.
  -UMSARS(Unified Multiple System Atrophy rating scale)
  The scale comprises the following components:
  Part I, historical, 12 items; Part II, motor examination, 14 items; Part III, autonomic examination; and Part IV, global disability scale (total UMSARS with scores ranging from 1 to 109)
  -K-MMSE(Korea Mini-Mental Status Examination)
  The scale comprises the following components:
  Orientation, memory, attention and calculation, naming and language, and drawing (total K-MMSE score of 30)
  -DSM-Ⅳ(Diagnostic and Statistical Manual of Mental Disorders)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Hyu Lee, MD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corestem Inc. — http://corestem.com/
- See also: Severance hospital Institutional Review Board — http://mdctc.yuhs.ac/HPC/Sinchon/IRB/IrbIntro